CLINICAL TRIAL: NCT02227173
Title: Effect of BMS-986020 on the Pharmacokinetics of Montelukast, Flurbiprofen, and Digoxin as Probe Substrates for CYP2C8, CYP2C9, and P-gp
Brief Title: A Phase 1 Drug-drug Interaction Study in Healthy Volunteers
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: IM136-004
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-10

CONDITIONS: Drug-drug Interaction Study
MeSH Terms: interventions — montelukast; Flurbiprofen; Digoxin

ARMS (1):
- Single-Sequence, A B C (Experimental): Treatment A:
  Single oral dose of montelukast, flurbiprofen, and digoxin on Day 1
  Treatment B:
  BMS-986020 orally twice daily (BID) on Day 8 through Day 10
  Treatment C:
  BMS-986020 orally BID, single oral dose of montelukast, flurbiprofen, and digoxin on Day 11; BMS-986020 BID on Day 12 through Day 17
  Interventions: Drug: BMS-986020; Drug: Montelukast; Drug: Flurbiprofen; Drug: Digoxin

INTERVENTIONS:
Drug: BMS-986020
Drug: Montelukast
Drug: Flurbiprofen
Drug: Digoxin

SUMMARY:
This is an open-label, single-sequence, drug-drug interaction study in healthy male and female subjects. There is no formal research hypothesis to be statistically tested. It is expected that coadministration of BMS-986020 with montelukast, flurbiprofen, and digoxin may increase the exposure of montelukast, flurbiprofen, and digoxin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female nonsmoking subjects ages 18 to 50 years, inclusive, with a body mass index of 18.0 to 32.0 kg/m2, inclusive
* Women of childbearing potential must agree to follow instructions for methods of contraception for the duration of the study

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of arrhythmias or palpitations associated with dizziness or fainting
* History of clinically relevant cardiac disease

Other protocol defined exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters (maximum observed plasma concentration, area under the concentration-time curve) for montelukast, flurbiprofen, and digoxin | Predose and up to 168 hours post dose
  Pharmacokinetic endpoints for montelukast, flurbiprofen, and digoxin with and without BMS-986020

SECONDARY OUTCOMES:
Additional pharmacokinetic parameters for montelukast, flurbiprofen, and digoxin. | Predose and up to 168 hour post dose
  Additional pharmacokinetic parameters for montelukast, flurbiprofen, digoxin, and with and without BMS-986020
Safety | From dosing (Day 1) to Day 21
  Collection of adverse events and other physical parameters to assess safety

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel DeNoia, MD, Principal Investigator — ICON Development Solutions
Locations (1):
- Healthcare Discoveries, LLC d/b/a ICON Development Solutions, San Antonio, Texas, United States